CLINICAL TRIAL: NCT06949072
Title: A Randomized, Single-Blind, Cross-Over Clinical Study to Assess an Experimental Dentifrice in an in Situ Model of Early Stage Caries
Brief Title: A Clinical Study to Assess an Experimental Dentifrice in an Experimental Model of Early Stage Caries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HALEON (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 300267
Record Dates: First submitted 2025-04-22; First posted 2025-04-29 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Dental Caries
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Test Dentifrice (Experimental): Participants will be instructed to dose the toothbrush provided with a strip of test dentifrice (a full brush head) and brush for one timed minute, twice daily (morning and evening) per the Brushing Instructions for up to 14 days each in Treatment Periods 1 to 3 as per crossover assignment. There will be a washout period of 2-3 days prior to each treatment period during which the participants will brush their teeth with the washout dentifrice for one timed minute, twice daily (morning and evening) per the Brushing Instructions.
  Interventions: Drug: Test Dentifrice
- Reference Dentifrice (Active Comparator): Participants will be instructed to dose the toothbrush provided with a strip of reference dentifrice (a full brush head) and brush for one timed minute, twice daily (morning and evening) per the Brushing Instructions for up to 14 days each in Treatment Periods 1 to 3 as per crossover assignment. There will be a washout period of 2-3 days prior to each treatment period during which the participants will brush their teeth with the washout dentifrice for one timed minute, twice daily (morning and evening) per the Brushing Instructions.
  Interventions: Drug: Reference Dentifrice
- Negative Control Dentifrice (Active Comparator): Participants will be instructed to dose the toothbrush provided with a strip of negative control dentifrice (a full brush head) and brush for one timed minute, twice daily (morning and evening) per the Brushing Instructions for up to 14 days each in Treatment Periods 1 to 3 as per crossover assignment. There will be a washout period of 2-3 days prior to each treatment period during which the participants will brush their teeth with the washout dentifrice for one timed minute, twice daily (morning and evening) per the Brushing Instructions.
  Interventions: Drug: Negative Control Dentifrice

INTERVENTIONS:
Drug: Test Dentifrice — Dentifrice containing 5 percent (%) weight by weight (w/w) Potassium nitrate (KNO3) and 1150ppm fluoride as sodium fluoride.
  Arms: Test Dentifrice
Drug: Reference Dentifrice — Dentifrice containing 1100ppm fluoride as stannous fluoride.
  Arms: Reference Dentifrice
Drug: Negative Control Dentifrice — Dentifrice containing 5% KNO3 with no fluoride.
  Arms: Negative Control Dentifrice

SUMMARY:
The aim of this study is to evaluate the relative efficacy of an experimental dentifrice containing 1150 parts per million (ppm) fluoride (as sodium fluoride [NaF]) to remineralize early stage caries type lesions in an in situ model compared to a negative control and a reference dentifrice.

DETAILED DESCRIPTION:
This is a randomized, single-blind, single-center, controlled, three period, three treatment, cross-over caries in situ model in healthy participants who wear a suitable removable mandibular partial denture. The denture will be modified to accommodate 2 gauze-covered, 4 millimeter (mm) round specimens of bovine dental enamel that have been previously demineralized in vitro to form artificial caries lesions. After 14 days of twice daily product use off-site, the specimens will be removed at the study site to determine the remineralization ability of the treatments. The same procedure will be followed for period 2 and 3 with a washout period of 2-3 days prior to each treatment period. Sufficient participants will be screened to randomize up to 50 participants to the study.

ELIGIBILITY:
Inclusion Criteria:

* Participant provision of a signed and dated informed consent document indicating that the participant has been informed of all pertinent aspects of the study before any assessment is performed.
* Participant is of either sex and any gender who, at the time of screening, is between the ages of 18-85 years, inclusive.
* Participant is willing and able to comply with scheduled visits, and other study procedures and restrictions.
* Participant is in good general and mental health with, in the opinion of the investigator or medically qualified designee, no clinically significant or relevant abnormalities in medical history or upon oral examination, or condition, that would impact the participant's safety, wellbeing or the outcome of the study, if they were to participate in the study, or affect the individual's ability to understand and follow study procedures and requirements.
* Participant who demonstrates a salivary flow-rate in the range of normal values (unstimulated whole saliva flow-rate more than or equal to (>=) 0.2 grams per minute (g/min); gum base stimulated whole saliva flow-Rate >= 0.8 g/min).
* Participant with a removable partial denture (RPD) fulfilling:

  1. Wears a removable mandibular partial denture that has good stability and support, with sufficient room on one side in the posterior teeth/buccal flange area to accommodate two enamel specimens (required dimensions approximately 5mm in diameter and 2.5mm deep for each specimen site).
  2. Willing to have their denture modified to accommodate the enamel test specimens.
  3. Willing and capable of wearing their removable partial dentures 24 hours per day during each 14-day treatment period.
  4. Willing and capable of brushing their natural teeth with the lower partial denture in place.
  5. Willing to cease using all denture cleaners and fixatives on their mandibular RPD during the study (with the exception of the supplied non-zinc fixative which may be used on any maxillary denture if present and required).

Exclusion Criteria:

* Participant who is an employee of the investigational site, either directly involved in the conduct of the study or a member of their immediate family; or an employee of the investigational site otherwise supervised by the investigator; or, a Haleon employee directly involved in the conduct of the study or a member of their immediate family.
* Participant who has participated in other studies (including non-medicinal studies) involving investigational product(s) within 30 days prior to study entry and/or during study participation.
* Participant with, in the opinion of the investigator or medically qualified designee, an acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator or medically qualified designee, would make the participant inappropriate for entry into this study.
* Participant who is pregnant (self-reported) or intending to become pregnant over the duration of the study or who is breastfeeding.
* Participant with known or suspected intolerance or hypersensitivity to the study materials (or closely related compounds) or any of their stated ingredients.
* Participant who, in the opinion of the investigator or medically qualified designee, has a condition or medical history that would impact on their safety or wellbeing or affect their ability to understand and follow study procedures and requirements or who should not participate in the study for other reasons.
* Participant with a recent history (within the last year) of alcohol or other substance abuse.
* Participant requiring the need for antibiotic premedication prior to a dental prophylaxis or taking some blood thinning medications that prohibit the safe conduct of a dental cleaning. Note: Medical consultation may need to be obtained from participant's physician at the examiner's discretion.
* Participant who is:

  1. Taking antibiotics or has taken antibiotics in the two weeks prior to the screening visit.
  2. Taking or has ever taken a bisphosphonate drug (that is, Fosamax, Actonel Boniva, Reclast, or Zometa).
  3. Using or intending to use professionally recommended fluoride supplements or fluoride mouth rinse, or has received a professional fluoride application in the 2 weeks prior to screening.
* Participant who has:

  1. Dental restorations in a poor state of repair that could impact participant safety or efficacy evaluations.
  2. Active caries or moderate or severe periodontal disease that may compromise the study or health of the participant. Participants presenting at screening with minor caries may continue in the study if their carious lesions are repaired prior to the start of the first treatment period.
* Participant who has previously been enrolled in this study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2025-04-28 (Actual); Primary Completion 2025-09-11 (Actual); Study Completion 2025-09-11 (Actual)

PRIMARY OUTCOMES:
Percent Surface Microhardness Recovery (%SMHr) After 2 Weeks in situ (Experimental Dentifrice Versus [Vs] Negative Control Dentifrice) | After 2 Weeks in situ in each Treatment Period
  The Surface Microhardness (SMH) technique is used to detect changes in the mineral content of dental enamel. The %SMHr will be derived as [(D1-R)/(D1-B)]*100, where D1= mean of replicate indentation lengths (micrometer [μm]) in enamel after first in vitro demineralization, R= mean of replicate indentation lengths (μm) in enamel after 2-weeks in situ and B= mean of replicate indentation lengths (μm) in sound enamel at baseline.

SECONDARY OUTCOMES:
%SMHr After 2 Weeks in situ (Experimental Dentifrice Vs Reference Dentifrice) | After 2 Weeks in situ in each Treatment Period
  The SMH technique is used to detect changes in the mineral content of dental enamel. The %SMHr will be derived as [(D1-R)/(D1-B)]*100, where D1= mean of replicate indentation lengths (μm) in enamel after first in vitro demineralization, R= mean of replicate indentation lengths (μm) in enamel after 2-weeks in situ and B= mean of replicate indentation lengths (μm) in sound enamel at baseline.
%SMHr After 2 Weeks in situ (Reference Dentifrice Vs Negative Control Dentifrice) | After 2 Weeks in situ in each Treatment Period
  The SMH technique is used to detect changes in the mineral content of dental enamel. The %SMHr will be derived as [(D1-R)/(D1-B)]*100, where D1= mean of replicate indentation lengths (μm) in enamel after first in vitro demineralization, R= mean of replicate indentation lengths (μm) in enamel after 2-weeks in situ and B= mean of replicate indentation lengths (μm) in sound enamel at baseline.
Transverse Microradiography (TMR) Parameter - Integrated Mineral Loss (∆Z) After 2 Weeks in situ | After 2 Weeks in situ in each Treatment Period
  Integrated Mineral Loss will be determined using TMR. TMR measures changes in mineral content by cutting the enamel specimens into plano-parallel thin slices and taking digitized microradiographic images of each. The mineral content is calculated from the gray intensity levels of the images of section.
TMR Parameter - Lesion Depth (L) After 2 Weeks in situ | After 2 Weeks in situ in each Treatment Period
  Lesion depth will be determined using TMR. TMR measures changes in mineral content by cutting the enamel specimens into plano-parallel thin slices and taking digitized microradiographic images of each. The mineral content is calculated from the gray intensity levels of the images of section.
TMR Parameter - Maximum Mineral Density at the Surface Zone (SZmax) After 2 Weeks in situ | After 2 Weeks in situ in each Treatment Period
  Maximum mineral density at the surface zone will be determined using TMR. TMR measures changes in mineral content by cutting the enamel specimens into plano-parallel thin slices and taking digitized microradiographic images of each. The mineral content is calculated from the gray intensity levels of the images of section.
Enamel Fluoride Uptake (EFU) After 2 Weeks in situ | After 2 Weeks in situ in each Treatment Period
  EFU gives valuable information regarding how much fluoride is incorporated into a remineralized lesion. In this technique the enamel is sampled through use of a microdrill to obtain a quantity of powdered enamel representative of the cross section through the lesion. The powder is dissolved in acid and chemically analyzed for fluoride.
Percent Net Acid Resistance (%NAR) After 2 Weeks in situ and Further in vitro Demineralization | After 2 Weeks in situ in each Treatment Period
  The resistance to acid-induced demineralization will be assessed through NAR. The %NAR (at the specimen level) will be derived as [(D1-D2)/(D1-B)]*100, where D1= mean of replicate indentation lengths (μm) in enamel after first in vitro demineralization, D2= mean of replicate indentation lengths (μm) in enamel after the second in vitro demineralization and B= mean of replicate indentation lengths (μm) in sound enamel at baseline.
Acid Resistance Ratio (ARR) After 2 Weeks in situ and Further in vitro Demineralization | After 2 Weeks in situ in each Treatment Period
  The resistance to acid-induced demineralization will be assessed through ARR. The ARR will be derived as 1-[(D2-R)/(D1-B)] where, D2= mean of replicate indentation lengths (μm) in enamel after the second in vitro demineralization, R= mean of replicate indentation lengths (μm) in enamel after 2-weeks in situ, D1= mean of replicate indentation lengths (μm) in enamel after first in vitro demineralization and B= mean of replicate indentation lengths (μm) in sound enamel at baseline.

CONTACTS AND LOCATIONS:
Locations (1):
- Oral Health Research Institute, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual participant data and study documents can be requested for further research from ww.clinical-trial-register@haleon.com
Supporting Information: Study Protocol, SAP, ICF
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months, but an extension can be granted, when justified, for up to another 12 months.